CLINICAL TRIAL: NCT00383786
Title: Evaluation of the Efficacy of the NK1 Antagonist GR205171 in Posttraumatic Stress Disorder
Brief Title: Substance P Antagonist in the Treatment of Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Sanjay Johan Mathew, MD, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 060253; 06-M-0253; NCT00211861 (obsolete NCT alias)
Record Dates: First submitted 2006-10-03; First posted 2006-10-04 (Estimated); Results first posted 2014-01-31 (Estimated); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: PTSD
Keywords: PTSD; Substance P; Treatment Study; Placebo; Controlled; Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — vofopitant; Psychophysiology; Spinal Puncture

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GR205171 (Experimental): selective neurokinin-1 receptor antagonist, fixed 5 mg dose every day, for 8 weeks.
  Interventions: Drug: NK1 Antagoist (GR205171); Procedure: Psychophysiology (Trauma Script); Procedure: Psychophysiology (Verbal Threat); Procedure: Psychophysiology (Fear Conditioning); Procedure: Psychophysiology (Affective Modulation); Procedure: Psychophysiology (Heart rate variability); Procedure: Lumbar Puncture; Procedure: 24-hour plasma sampling; Procedure: MRI
- placebo (Placebo Comparator): sugar pill
  Interventions: Procedure: Psychophysiology (Trauma Script); Procedure: Psychophysiology (Verbal Threat); Procedure: Psychophysiology (Fear Conditioning); Procedure: Psychophysiology (Affective Modulation); Procedure: Psychophysiology (Heart rate variability); Procedure: Lumbar Puncture; Procedure: 24-hour plasma sampling; Procedure: MRI

INTERVENTIONS:
Drug: NK1 Antagoist (GR205171)
  Arms: GR205171
Procedure: Psychophysiology (Trauma Script)
Procedure: Psychophysiology (Verbal Threat)
Procedure: Psychophysiology (Fear Conditioning)
Procedure: Psychophysiology (Affective Modulation)
Procedure: Psychophysiology (Heart rate variability)
Procedure: Lumbar Puncture
Procedure: 24-hour plasma sampling
Procedure: MRI

SUMMARY:
This study, conducted at the NIH and the Mount Sinai School of Medicine, will examine the effectiveness of a substance P or NK1 antagonist study drug known as GR205171 in treating the symptoms of posttraumatic stress disorder (PTSD).

People between 18 and 65 years of age who have been diagnosed with PTSD may be eligible for this study. Participants undergo the following tests and procedures:

Treatment: Patients are tapered off current ineffective medications over 1 to 2 weeks. All participants receive placebo (sugar pill) at the start of the study. At some point within the first 3 weeks of the study, they are then randomly assigned either to take GR205171 or to continue with placebo for the remainder of the 10-week treatment period.

Clinic visits: Patients come to the clinic once a week during treatment. The following procedures are done at various visits.

* Interviews, self report questionnaires and psychiatric rating scales at every visit.
* Physical examination, blood and urine tests. Blood is drawn up to 10 times during the study.

Follow-up visits continue for up to 3 months after the end of the study, during which patients are offered standard clinical treatment.

DETAILED DESCRIPTION:
Posttraumatic Stress Disorder (PTSD) is a common chronic anxiety disorder that is often debilitating and follows exposure to an overwhelming traumatic event. The burden of PTSD on individuals and society is significant. The majority of PTSD sufferers also meet the diagnostic criteria for several other psychiatric disorders and many attempt suicide. Despite the devastating impact of PTSD on the lives of millions worldwide, little is known about the etiology or pathophysiology of this disorder. Although disruptions in the hypothalamic-pituitary adrenal (HPA) Axis, noradrenergic, serotonergic systems have been proposed as neurobiological substrates in the development of PTSD, the exact underpinnings of the neurobiology of PTSD remain to be fully elucidated.

PTSD is responsive to treatment with selective serotonin reuptake inhibitors, but response rates rarely exceed 60%, and even fewer patients (20%-30%) experience improvement that could be characterized as remission. Thus, there is a clear need to develop novel and improved therapeutics for PTSD. A growing body of preclinical evidence suggests that activation of the Substance P (SP) and its receptor NK1 is anxiogenic and that NK1 antagonists, upon chronic administration, exert significant dampening (albeit complex) effects on the SP-NP system. Furthermore, several stress paradigms are believed to exert many of their deleterious effects on hippocampal structures via enhancement of SP-NK1 system. Overall, excess activity of the SP-NK1 system stands as a prime candidate for involvement in the pathophysiology of anxiety disorders such as PTSD.

In this study, we propose to investigate the potential antianxiety efficacy of the highly specific NK1 antagonist GR205171 in PTSD. Furthermore, we propose to, in a preliminary fashion, longitudinally investigate whether neuroendocrine surrogate markers are predictive of treatment response.

This is an 8-week double-blind placebo-controlled study that will examine the efficacy and safety of an NK1 antagonist in patients with PTSD.

Patients, ages 18 to 65 years with a diagnosis of PTSD, will in this pilot study be randomized to double-blind treatment to receive either the NK1 antagonist, GR205171 (5 mg/day) or placebo for a period of 8 weeks.

Approximately 52 patients will enter the study to obtain 40 subjects who complete the 8 weeks of acute NK1 antagonist treatment.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects may be included in the study only if they meet all of the following criteria:

1. Male or female subjects, 18 to 65 years.
2. Female subjects of childbearing potential must be using a medically accepted means of contraception.
3. Each subject must have a level of understanding sufficient to agree to all required tests and examinations and sign an informed consent document.
4. A negative urine toxicology.
5. Subjects must fulfill the criteria for PTSD as defined in DSM-IV (309.81), which should be the primary diagnosis. Diagnoses are based on clinical assessment and confirmed by structured diagnostic interview SCID-P.
6. Duration of illness of PTSD for at least 3 months.
7. Subjects must have an initial score at Visit 1 and Visit 2 of at least 50 on the CAPS for PTSD Studies.
8. Subjects must not have a decrease in the total score of CAPS of greater than 25% during washout (between Visits 1 and 2).

EXCLUSION CRITERIA:

Subjects will be excluded from the study for any of the following reasons:

1. Presence of psychotic features.
2. Participation in a clinical trial of another investigational drug within 1 month (30 days) prior to study entry (Visit 1).
3. Female subjects who are either pregnant or nursing.
4. Serious, unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease.
5. Subjects with uncorrected hypothyroidism or hyperthyroidism.
6. Previous treatment with NK1 receptor antagonist.
7. DSM-IV substance abuse or dependence within the past 90 days.
8. Treatment with an injectable depot neuroleptic within less than one dosing interval between depot neuroleptic injections prior to Visit 2.
9. Treatment with a reversible MAOI, guanethidine, or guanadrel within 1 week or with fluoxetine within 6 weeks prior to Visit 2.
10. Treatment with any other concomitant medication with primarily CNS activity.
11. Treatment with clozapine or ECT within 12 weeks prior to Visit 2.
12. Current diagnosis of schizophrenia or other psychotic disorder, bipolar disorder, other Axis I disorder (except for major depressive disorder, dysthymia and other anxiety disorders that followed exposure to the trauma) as defined in the DSM-IV.
13. Patients who are currently at high risk for homicide or suicide, a score greater than 4 on item 10 of the MADRS.
14. Current or planned litigation regarding the traumatic event.

Patients will not be allowed to receive structured psychotherapy during the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis S Charney, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Mt. Sinai Medical Center, New York, New York

REFERENCES:
- [Background] Agelink MW, Boz C, Ullrich H, Andrich J. Relationship between major depression and heart rate variability. Clinical consequences and implications for antidepressive treatment. Psychiatry Res. 2002 Dec 15;113(1-2):139-49. doi: 10.1016/s0165-1781(02)00225-1. PMID 12467953
- [Background] Ballard TM, Sanger S, Higgins GA. Inhibition of shock-induced foot tapping behaviour in the gerbil by a tachykinin NK1 receptor antagonist. Eur J Pharmacol. 2001 Feb 2;412(3):255-64. doi: 10.1016/s0014-2999(01)00724-5. PMID 11166289
- [Background] Bernstein EM, Putnam FW. Development, reliability, and validity of a dissociation scale. J Nerv Ment Dis. 1986 Dec;174(12):727-35. doi: 10.1097/00005053-198612000-00004. PMID 3783140
- [Derived] Mathew SJ, Vythilingam M, Murrough JW, Zarate CA Jr, Feder A, Luckenbaugh DA, Kinkead B, Parides MK, Trist DG, Bani MS, Bettica PU, Ratti EM, Charney DS. A selective neurokinin-1 receptor antagonist in chronic PTSD: a randomized, double-blind, placebo-controlled, proof-of-concept trial. Eur Neuropsychopharmacol. 2011 Mar;21(3):221-9. doi: 10.1016/j.euroneuro.2010.11.012. Epub 2010 Dec 30. PMID 21194898

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients (aged 18-65) were recruited from media advertisement (86%) or clinician referral (14%). Diagnoses were made with the SCID-IV performed by an experienced research clinician, along with an independent interview by a psychiatrist. A primary diagnosis of chronic PTSD, signifying an illness duration.
Pre-assignment Details: Of 235 potential participants screened for eligibility, 171 (73%) were excluded prior to placebo lead-in. 128 did not meet eligibility criteria, 24 were lost to follow-up, and 19 withdrew consent. Sixty-four patients began placebo lead-in, of whom 47 patients (73%) were randomized (11 were ineligible and 6 withdrew consent).
Groups:
- GR205171: selective neurokinin-1 receptor antagonist, 5mg/day for a period of 8 weeks
- Placebo: sugar pill administered daily for a period of 8 weeks
Period: Overall Study
Arm/Group | GR205171 | Placebo
Started | 22 | 25
Completed | 18 | 13
Not Completed | 4 | 12
Not completed — Protocol Violation | 2 | 6
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- GR205171: selective neurokinin-1 receptor antagonist
- Total: Total of all reporting groups
Arm/Group | GR205171 | Placebo | Total
Number analyzed (Participants) | 22 | 25 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 25 | 47
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (11.5) | 38.7 (12.3) | 40.9 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 23
  Male | 10 | 14 | 24
Region of Enrollment [Number; unit: participants]
  United States | 22 | 25 | 47

OUTCOME MEASURES:

1. Primary Outcome: Changes in CAPS Scores.
Description: The Clinician-Administered PTSD Scale (CAPS) is the gold standard in PTSD assessment. The CAPS is a 30-item structured interview that corresponds to the DSM-IV criteria for PTSD. This is a 17-item core symptom scale, measuring both frequency and intensity of symptoms, with the most frequently used scoring rule is to count a symptom as present if it has a frequency of 1 or more and an intensity of 2 or more. A PTSD diagnosis is made if there is at least 1 "B" symptom, 3 "C" symptoms, and 2 "D" symptoms as well as meeting the other diagnostic criteria. Scores range from 0-136 0 (best possible outcome) to 136 (worst possible outcome). The relevant time-points for reporting change were at baseline and 8 weeks.
Time Frame: Baseline, 8 weeks
Population: 20 patients randomized to drug were included in the primary analysis as 2 our of the 22 randomized were excluded because they did not receive a week 1 assessment. 19/25 randomized to placebo were included in the analysis after 6 were excluded due to not receiving week 1 assessments.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | GR205171 | Placebo
Number analyzed (Participants) | 20 | 19
scores on a scale | 43.5 (5.1) | 51.1 (5.7)

2. Other Pre Specified Outcome: Able to Identify Biological Markers That Predict Response to Treatment.
Time Frame: 10 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | GR205171 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/25
Other Adverse Events (participants affected / at risk) | 13/22 | 6/25
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GR205171 (N=22) | Placebo (N=25)
Headache (Nervous system disorders) | 13 | 6

LIMITATIONS AND CAVEATS:
Limitations include the small sample size and brief duration of the trial, as 8 weeks might have been insufficient to test the efficacy of GR205171 for chronic PTSD. Sample size was also a limitation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No